CLINICAL TRIAL: NCT03758001
Title: Phase Ia/Ib Trial to Evaluate the Tolerability and Safety of IBI101 Monotherapy or in Combination With Sintilimab in Advanced Solid Tumor Patients
Brief Title: First in Human Study of IBI101 in Chinese Subjects With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CIBI101A101
Record Dates: First submitted 2018-11-01; First posted 2018-11-29 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IBI101 (Experimental): IBI101 will be administrated intravenously. 3+3 dose escalation design will be used with eight dose levels being tested.
  Interventions: Drug: IBI101
- IBI101 in combination with Sintilimab (Experimental): IBI101 and Sintilimab will be administrated intravenously. 3+3 dose escalation design will be used with 4 dose levels of IBI101 being tested.
  Two dose levels of IBI101 in combination with Sintilimab will be expanded to 10 patients each.
  Interventions: Drug: IBI101; Drug: Sintilimab

INTERVENTIONS:
Drug: IBI101 — 0.01 mg/kg; 0.1 mg/kg; 0.3 mg/kg; 1 mg/kg; 3 mg/kg; 6 mg/kg; 10 mg/kg; 15 mg/kg iv infusion day 1 of every 21 days
  Arms: IBI101
Drug: IBI101 — 1 mg/kg; 3 mg/kg; 6 mg/kg; 10 mg/kg iv infusion day 1 of every 21 days
  Arms: IBI101 in combination with Sintilimab
Drug: Sintilimab — 200mg iv infusion day 1 of every 21 days
  Other Names: IBI308
  Arms: IBI101 in combination with Sintilimab

SUMMARY:
Phase 1a/1b Trial to evaluate the tolerability and safety of IBI101 monotherapy or in combination with Sintilimab in advanced solid tumor patients.

DETAILED DESCRIPTION:
IBI101 and Sintilimab will be administered intravenously on Day 1 of every 21-day cycle. The DLT observation period is 21 days starting with the first dose taken on day 1. In the Phase Ia study, eight dose levels of IBI101 (0.01, 0.1, 0.3, 1, 3, 6, 10 and 15mg/kg) will be tested. In the Phase Ib study, four dose levels of IBI101 (1, 3, 6 and 10mg/kg), in combination with Sintilimab 200mg, will be tested. After completion of the dose escalation phase, two combination dose cohorts (IBI101 3mg/kg and 6mg/kg, in combination with Sintilimab 200mg) will be expanded to 10 patients each.

IBI101 is a recombinant fully humanized IgG1 anti-tumor necrosis factor receptor superfamily member 4 (OX40) monoclonal antibody.

Sintilimab is a recombinant fully humanized anti-programmed death 1 (PD1) monoclonal antibody.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced, recurrent or metastatic solid tumors who have failed standard treatment
* 18 to 75 years old
* Life expectancy ≥ 12 weeks
* At least 1 measurable lesion
* ECOG PS score 0 or 1
* Adequate organ and bone marrow function

Exclusion Criteria:

* Previous exposure to anti-OX40, anti-PD-1, anti-PD-L1, anti-PD-L2 antibody or other immune checkpoint inhibitors
* Exposure to any other investigational drug in the 4 weeks prior to 1st dose of investigational drug
* Exposure to anti-tumor agents in the 3 weeks prior to 1st dose of investigational drug
* Exposure to immunosuppressant in the 3 weeks prior to 1st dose of investigational drug
* Major surgery in the 4 weeks prior to 1st dose of investigational drug
* 30Gy radiation in the chest in the 6 months prior to 1st dose of investigational drug
* History of autoimmune disease
* Symptomatic CNS metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-02-13 (Actual); Primary Completion 2023-02-16 (Actual); Study Completion 2023-02-16 (Actual)

PRIMARY OUTCOMES:
Incicende of Adverse Events (AEs) | 2 years
  Number of patients with AE, treatment-related AE (TRAE), immune-related AEs (irAE), AE of special interest (AESI), serious adverse event (SAE), discontinuation of study drug due to AE, dose-limiting toxicity (DLT) assessed by CTCAE v5.0.

SECONDARY OUTCOMES:
Overall response rate (ORR) | 2 years
Time to response (TTR) | 2 years
Duration of response (DOR) | 2 years
Progression free survival (PFS) | 2 years
Area Under Curve (AUC)last and AUC0-inf | 2 years
Maximum Concentration (Cmax) | 2 years
Total body clearance (CL) | 2 years
Volume of distribution (Vz) | 2 years
Time at which maximum concentration occurred (Tmax) | 2 years
Elimination half-life (t1/2) | 2 years
Mean residue time (MRT) | 2 years
OX40 receptor occupancy | 2 years
T cell subset analysis | 2 years
Anti-drug antibody (ADA) | 2 years
Neutralizing antibody (Nab) positive rate | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China